CLINICAL TRIAL: NCT00515918
Title: The Effect of Early Iron Deficiency on Developmental Brain and Behavior in Infants
Acronym: IDBB
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Other Study IDs: C030104-30671773
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2007-08-14 (Estimated); Status verified 2007-08

CONDITIONS: Iron Deficiency
Keywords: Iron deficiency; brain; cognition; behavior
MeSH Terms: conditions — Iron Deficiencies; Behavior | interventions — Iron

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Iron deficient
  Interventions: Dietary Supplement: iron
- 2: Iron sufficient

INTERVENTIONS:
Dietary Supplement: iron
  Groups: 1

SUMMARY:
The purpose of this project to examine brain functions and behavior related to ID including sensory ,motor, cognitive and social /emotional functioning, and address unanswered questions about brain and behavior impacts of different timing of ID(pre- and /or postnatal ID) in infants.

DETAILED DESCRIPTION:
Iron deficiency (ID) is the most common single nutrient disorder in the world. Pregnant women and children before pre-school age are at highest risk. Data from animal models provide evidence that early ID affected developing brain in specific regions and functions by varies processes include myelination, dopamine neurotransmitter system, and neurometabolism. These impacts appeared differential at different time of brain development and different brain regions, depending on the timing of ID. The reversibility of these effects also appeared to depend on the timing of ID. This project uses innovative neuropsychologic/ neurophysiologic and behavioral techniques, such as event-related potentials(ERP), ABR and VEP, to study brain functions and behavior related to ID including sensory ,motor, cognitive and social /emotional functioning, and address unanswered questions about brain and behavior impacts of different timing of ID(pre- and /or postnatal ID) in the human infants. This research has the potential to understand reversibility of effects depending on timing of ID and treatment as well as basic understanding of mechanism of impact of ID in human developing brain. It may also have important implications with regard to policy of interventions for different timing of ID, and improve children early development and the quality of population.

ELIGIBILITY:
Inclusion Criteria:

* Full- term infants

Exclusion Criteria:

* Prematures,
* Perinatal high risk infants(asphyxia,infection etc.),
* Maternal alcohol,
* Smoking,
* Drug abuse,
* Inherited diseases

Max Age: 36 Months | Sex: All
Age Groups: Child
Dates: Start 2007-09; Study Completion 2010-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Zhengyan Zhao, M.D, Principal Investigator — Zhejiang University School of Medicine, Children's Hosp
Locations (1):
- Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China